CLINICAL TRIAL: NCT05074290
Title: Pharmacokinetics and Safety of Epidiferphane and Taxanes in Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UF-BRE-007
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; taxanes; Epidiferphane
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epidiferphane + taxane chemotherapy (Experimental)
  Interventions: Drug: Epidiferphane; Drug: Taxane Chemotherapy

INTERVENTIONS:
Drug: Epidiferphane — During the phase I portion of the study, subjects will be assigned to take either two (half target dose) or four (full target dose) Epidiferphane tablets orally three times daily following a 3 + 3 design. Three subjects will be sequentially enrolled at each of the 2 dose levels (beginning with the half target dose) until at least one dose-limiting toxicity (DLT) occurs. Dosing escalation will be stopped if two or more DLTs occur at either dose level. The maximum tolerated dose will be one dose level lower than the dose level at which 2 or more DLTs occur. Dose escalation will occur separately for each taxane regimen (docetaxel or paclitaxel).
  All subjects in the phase II portion of the study will receive the maximum tolerated dose determined in the phase I portion of the study for their taxane regimen.
  Subjects in both portions of the study will receive treatment with Epidiferphane for a maximum of three months.
Drug: Taxane Chemotherapy — All subjects on both phases of the study will be concurrently treated with a taxane regimen containing either paclitaxel given weekly, nab-paclitaxel given weekly or every 3 weeks or docetaxel given every 3 weeks. The choice of taxane regimen will be determined by the treating physician prior to consenting to participate in this trial.

SUMMARY:
Patients with breast cancer are commonly treated with taxane chemotherapy. Some very common side effects of taxanes, such as anemia and peripheral neuropathy, are often as not well addressed during treatment, resulting in dose reductions, dose delays and early discontinuation (collectively called relative dose intensity) of these chemotherapy agents in 15-80 % of patients on these drugs. This reduction in relative dose intensity (RDI) results in worse clinical outcomes such as progression free and overall survival. Pre-clinical studies in mouse models subjected to standardized chemotherapy regimens containing paclitaxel or oxaliplatin have shown that the nutritional supplement Epidiferphane reduces both neuropathy and anemia. This study will investigate whether the use of Epidiferphane in patients with breast cancer receiving taxane chemotherapy results in an attenuation of the side effects experienced, as well as an improvement in tumor response rate. The safety and maximum tolerated dose of Epidiferphane in this patient population will also be determined in this study.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Subjects on the phase I portion must either be initiating neoadjuvant chemotherapy or have a clinical diagnosis of metastatic breast cancer. Subjects on the phase II portion must have a clinical diagnosis of breast cancer of any stage and histology.
* Must be about to start a new treatment regimen containing either paclitaxel given weekly or docetaxel given every 3 weeks or nab-paclitaxel given weekly or every 3 weeks at UF Health, at one of the following doses:

  * Paclitaxel weekly at 80-90 mg/m2
  * Nab-paclitaxel weekly at 75-125 mg/m2 or every three weekly at 260 mg/m2
  * Docetaxel every three weeks at 75-100 mg/m2
* An ECOG Performance Status less than or equal to 3 based on treating physician assessment
* Must continue cancer therapy at UF Health for at least the next three months
* Must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included.
* A functioning digestive tract with no obstruction
* Subjects must be willing to avoid regular consumption of green tea and curcumin supplements for the duration of trial participation.
* Written informed consent obtained from the subject and the ability for the subject to comply with all the study-related procedures.
* Subjects of childbearing potential (SOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study.
* Subjects with partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study.

Exclusion Criteria:

* Must not be receiving any other investigational agents
* Subjects of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and following completion of taxane therapy for an additional 6 months for subjects of child bearing potential and 3 months for subjects with partners of child bearing potential.
* Subjects who are pregnant or breastfeeding
* Active systemic infection considered to be opportunistic, life threatening or clinically significant at the time of treatment.
* Psychiatric illness or social situation that would limit compliance with trial requirements.
* Known allergy to turmeric, broccoli, or green tea.
* Subjects must not be on treatment with strong CYP3A4 inhibitors such as tacrolimus or on verapamil during the trial.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding (e.g. hemoglobin < 10 mg/dL, CTCAE v 5.0 grade 3 or higher neutropenia or thrombocytopenia) giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.
* CTCAE v 5.0 grade 2 or higher peripheral sensory or motor neuropathy
* CTCAE v 5.0 grade 1 or higher paresthesia
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >2.5 × the upper limit of normal (ULN)
* Total bilirubin (TBL) >1.5 × ULN or >3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia)
* Glomerular filtration rate (GFR) <50 mL/min
* Red blood cell infusions < 30 days prior to treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cmax of Epidiferphane's components | 24 hours
  The Cmax of each of Epidiferphane's components will be based on blood concentration measured prior to taxane chemotherapy administration, as well as at 1, 2 and 24 hours after taxane chemotherapy administration.
  The Cmax of each of Epidiferphane's components will be the blood concentration measured prior to taxane chemotherapy administration, as well as at 1, 2 and 24 hours after taxane chemotherapy administration.
Cmax of taxanes | 24 hours
  The Cmax of the taxane chemotherapy agents given will be based on blood concentrations measured prior to taxane chemotherapy administration, as well as at 1, 2 and 24 hours after taxane chemotherapy administration.
Concentration at 24 hours (C24 hours) of Epidiferphane's components | 24 hours
  The C24 hours of each of Epidiferphane's components will be based on blood concentration measured 24 hours after taxane chemotherapy administration.
Concentration at 24 hours (C24 hours) of taxanes | 24 hours
  The C24 hours of the taxanes given will be based on blood concentration measured 24 hours after taxane chemotherapy administration.
Maximum tolerated dose of Epidiferphane in patients with breast cancer who are being treated with taxanes | 4 months
Rate of Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade 2 or higher neuropathy | 4 months
Rate of Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade 1 or higher anemia | 4 months

SECONDARY OUTCOMES:
Effect of Epidiferphane on quality of life, as measured by the EORTC QLQ-C30 scale | 3 months
  The EORTC QLQ-C30 measures ability to perform everyday activities and whether the subject has experienced select physical symptoms on a scale of 1-4 (with 1 meaning "Not at all" and 4 meaning "Very much"), as well as overall quality of life and overall healt over the past week on a scale from 1-7 (with 1 meaning "Very Poor" and 7 meaning "Excellent").
Effect of Epidiferphane on quality of life, as measured by the FACT-Taxane scale | 3 months
  The FACT-Taxane measures various aspects of physical, social, emotional, and functional well-being, as well as whether the subject has experienced select physical symptoms over the past 7 days, on a scale of 0-4 (with 0 meaning "Not at all" and 4 meaning "Very much").
Objective response rate | 3 months
  Determine the objective response rate, defined as the percentage of subjects with a complete or partial response, as measured by RECIST 1.1 criteria, or descriptive statistics if RECIST measurements are not possible due to modality of imaging.
Concentration of the neuropathy marker NF-kB, as measured by multiplex cytokine bead analysis or ELISA (enzyme-linked immunosorbent assay) | 3 months
Concentration of the neuropathy marker VEGFA, as measured by multiplex cytokine bead analysis or ELISA (enzyme-linked immunosorbent assay) | 3 months
Concentration of the neuropathy marker Nrf2, as measured by multiplex cytokine bead analysis or ELISA (enzyme-linked immunosorbent assay) | 3 months
Concentration of the neuropathy marker IL18, as measured by multiplex cytokine bead analysis or ELISA (enzyme-linked immunosorbent assay) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Coy Heldermon, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States